CLINICAL TRIAL: NCT01196013
Title: A Phase I, Open-label, Multi-center Study of Clofarabine in Japanese Paediatric Patients With Relapsed or Refractory Acute Lymphoblastic Leukaemia
Brief Title: A Study of Clofarabine in Japanese Paediatric Patients With Relapsed or Refractory Acute Lymphoblastic Leukaemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLO05908
Record Dates: First submitted 2010-09-03; First posted 2010-09-08 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-03

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Clofarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Clofarabine (Experimental)
  Interventions: Drug: Clofarabine

INTERVENTIONS:
Drug: Clofarabine — Intravenous, 30 mg/m2, 52 mg/m2
  Other Names: Evoltra, Clolar, JC0707

SUMMARY:
The purpose of this study is primarily to assess the safety, tolerability and pharmacokinetics (PK) of clofarabine intravenously administered to pediatric patients with relapsed or refractory acute lymphoblastic leukemia (ALL) or for whom no other therapy with greater potential clinical benefit exists. The dosing regimen for the intravenous (IV) clofarabine is 30 or 52 mg/m2/day for 5 consecutive days. The secondary objectives are to document the activity of clofarabine and to explore the impact of deoxycytidine kinase (dCK) promoter polymorphism on PK and treatment outcome.

DETAILED DESCRIPTION:
This is a Phase I Study of Clofarabine in Japanese Paediatric Patients With Relapsed or Refractory Acute Lymphoblastic Leukaemia.

Subjects will receive intravenous administration of clofarabine at 30 or 52 mg/m2/day (2 hours) for 5 consecutive days and then the administration will be withheld until Day 14. If there is no evidence of recovery in neutrophil (≥750/mm3) and/or platelet count (≥50,000/mm3), the therapy may be withheld up to Day 42. However, in the absence of progression based on the judgment of the investigator after each cycle of treatment and the benefit of continued treatment is judged to exceed the risk, subjects may receive up to a total of six cycles. If a subject is receiving two or more cycles, a written consent must be obtained prior to start of Cycle 2.

When a subject completes the final dose, the safety will be observed and followed-up for 45 days after the final study drug administration.

Cohort 1 will receive 30 mg/m2/day x 5 days at Cycle 1 and will be assessed for tolerability. Samples will be drawn to assess pharmacokinetics at this dose. If subjects do not develop adverse events indicative of dose limiting toxicity (DLT) at Cycle 1, the dose will be increased to 52 mg/m2/day x 5 days from Cycle 2 and the subjects will be assessed for safety and activity only.

Cohort 2 will receive 52 mg/m2/day x 5 days at Cycle 1 and will be assessed for the tolerability. Samples will be drawn to assess pharmacokinetics at this dose.

Whether or not proceeding to Cohort 2 after the Cycle 1 of Cohort 1 is completed will be determined by the sponsor based on the assessment of the safety data and the recommendation of the Data Safety Monitoring Board (DSMB).

ELIGIBILITY:
Inclusion Criteria:

* Signed and written informed consent provided by patients ≥ 20 years old or by the parents or guardians of patients less than 20 years old. Investigator should verbally obtain informed assent from the patients 7 years old or older and written informed assent from patients 12 years old or older.
* Greater than or equal to 25 percent blasts present in the bone marrow and/or peripheral blood count and diagnosed with ALL .at time of enrollment
* Patients with relapsed or refractory ALL. Patients must not be eligible for therapy of higher clinical benefit potential and must be in second or subsequent relapse and/or refractory, i.e. failed to achieve remission following 2 or more different regimens, or for whom no other therapy with greater potential clinical benefit exists.
* Have a Karnofsky Performance Status of greater than or equal to 70 for patients 10 years of age or older or Lansky Performance Status greater than or equal to 70 for patients below 10 years of age.
* Patients whose hepatic, renal, and pancreatic functional tests are within the ranges defined in the protocol.

Exclusion Criteria:

* Received previous treatment with clofarabine.
* Have received any other investigational agent within 30 days prior to the first dose of the study drug.
* Have received any other chemotherapy within 14 days prior to the first dose of clofarabine. However, intrathecal drug administration is allowed up to 24 hours prior to the first dose of clofarabine. In addition, the patient must have been recovered from acute toxicity related to other chemotherapy or investigational agents (baseline or less than or equal to Common Terminology Criteria for Adverse Events ver 3.0 Grade 1)
* Have systemic fungal, bacterial, viral, or other infection that cannot be controlled(defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment). In addition, for patients with a history of fever (≥38.5˚C) within the preceding 3 days at the time of enrollment, documentation of negative blood cultures for at least 48 hours required.
* Have a psychiatric disorder that would interfere with consent, study participation, or follow-up.
* Patients whose spinal fluid tested immediately before the study registration within 7 days before dose indicates symptomatic Central Nervous System (CNS) involvement (i.e.CNS3).
* Have any other severe concurrent disease or a history of serious organ dysfunction or disease involving the heart, kidney, liver, or pancreas.
* Have received hematopoietic stem cell transplantation (HSCT) within 3 months prior to providing the consent or have acute graft-versus-host disease (GVHD) (greater than or equal to Grade 2) requiring immunosuppressive therapy or severe (systemic) chronic GVHD.
* Have a prior positive test for Hepatitis B surface (HBs) antigen or antibody, HBc antibody, Hepatitis C virus (HCV) antibody, or human immunodeficiency virus (HIV) antibody. (The patients who have had treatment of vaccine and are positive for HBs antibody are eligible).
* Are pregnant or nursing. Male and female patients of reproductive potential must agree to use an effective means of birth control to avoid pregnancy during the study period and for 180 days after the last dose of study drug.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2010-08; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 14 days (1st cycle)
Safety as evaluated by adverse events (incidence, severity, duration, causality, seriousness, type) | 45 days after final study drug administration
Pharmacokinetics as measured by maximum drug serum concentration (Cmax) | Day 1 to Day 5
Pharmacokinetics as measured by Time to maximum serum concentration (Tmax) | Day 1 to Day 5
Pharmacokinetics as measured by Area Under the drug-concentration curve (AUC) | Day 1 to Day 5
Pharmacokinetics as measured by half life (t1/2) | Day 1 to Day 5
Pharmacokinetics as measured by renal clearance (CLr) | Day 1 to Day 5

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (9):
- Japan (9):
  - National Kyusyu Cancer Center, Fukuoka
  - Fukushima Medical University Hospital, Fukushima
  - Kagoshima University Medical and Dental Hospital, Kagoshima
  - Tokai University Hospital, Kanagawa
  - Niigata Cancer Center Hospital, Niigata
  - Osaka City General Hospital, Osaka
  - Saitama Chilidren's Medical Center, Saitama
  - Shizuoka Children's Hospital, Shizuoka
  - St. Luke's International Hospital, Tokyo